CLINICAL TRIAL: NCT05660369
Title: INCIPIENT: INtraventricular CARv3-TEAM-E T Cells for PatIENTs With GBM
Brief Title: CARv3-TEAM-E T Cells in Glioblastoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Marcela V. Maus, M.D.,Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Marcela V. Maus, M.D.,Ph.D., Sponsor Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-175
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Glioblastoma; Malignant Glioma; Recurrent Glioblastoma; Recurrent Glioma
Keywords: Glioblastoma; Malignant Glioma; Recurrent Glioblastoma; Recurrent Glioma; Immunotherapy; Gene-Transfer Therapy
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Safety Run-In Phase (Experimental): * Participant enrollment will be staggered by 30 days for up to 3 participants.
  * Participants will receive 1 infusion of CARv3-TEAM-E.
  * Phase will be expanded up to 6 participants if any Dose-Limiting Toxicities DLTs occur.
  * After all participants have been enrolled, there will be an evaluation made by the Data Safety Monitoring Board (DSMB) and the FDA to determine the safety of enrollment into additional arms.
  Interventions: Drug: CARv3-TEAM-E T cells
- Arm 1: Recurrent Glioblastoma (GBM), EGFRvIII Positive (Experimental): * Participants will undergo a leukapheresis procedure, or collection of mononuclear T cells via peripheral blood draw.
  * Rituximab will be administered 5-10 days prior to infusion.
  * Lymphodepletion chemotherapy treatment will occur 5 days prior to infusion.
  * CARv3-TEAM-E will be administered via Ommaya on D0
  * Participants will be followed for 2 years post-treatment.
  * Participants who are deriving clinical benefit and have sufficient product can be retreated with up to 5 additional doses.
  Interventions: Drug: CARv3-TEAM-E T cells
- Arm 2: Newly Diagnosed GBM, EGFRvIII Positive (Experimental): * Participants will undergo a leukapheresis procedure, or collection of mononuclear T cells via peripheral blood draw.
  * Rituximab will be administered 5-10 days prior to infusion.
  * Lymphodepletion chemotherapy treatment will occur 5 days prior to infusion.
  * CARv3-TEAM-E will be administered via Ommaya on D0
  * Participants will be followed for 2 years post-treatment.
  * Participants who are deriving clinical benefit and have sufficient product can be retreated with up to 5 additional doses.
  Interventions: Drug: CARv3-TEAM-E T cells
- Arm 3: Recurrent GBM, EGFRvIII Negative (Experimental): * Participants will undergo a leukapheresis procedure, or collection of mononuclear T cells via peripheral blood draw.
  * Rituximab will be administered 5-10 days prior to infusion.
  * Lymphodepletion chemotherapy treatment will occur 5 days prior to infusion.
  * CARv3-TEAM-E will be administered via Ommaya on D0
  * Participants will be followed for 2 years post-treatment.
  * Participants who are deriving clinical benefit and have sufficient product can be retreated with up to 5 additional doses.
  Interventions: Drug: CARv3-TEAM-E T cells

INTERVENTIONS:
Drug: CARv3-TEAM-E T cells — Autologous T lymphocyte population that contains cells transduced ex-vivo with a CARv3-TEAM-E lentiviral vector encoding a chimeric antigen receptor (CAR). Administered via Ommaya reservoir.
  Other Names: Autologous T lymphocyte

SUMMARY:
The goal of this research study is to determine the best dose of CARv3-TEAM-E T Cells for treating participants with glioblastoma.

The name of the treatment intervention used in this research study is:

-CARv3-TEAM-E T Cells (or Autologous T lymphocytes).

DETAILED DESCRIPTION:
This is a non-randomized, open label, single site Phase 1 study to define the appropriate dose of CARv3-TEAM-E and evaluate its safety for the treatment of recurrent or newly diagnosed glioblastoma.

The U.S. Food and Drug Administration (FDA) has not approved CARv3-TEAM-E T Cells as a treatment for any disease. This is the first time that CARv3-TEAM-E T Cells will be given to humans. CARv3-TEAM-E T Cells are made from a person's own collected immune cells (T-Cells) that are genetically changed and then delivered back into the body to try to kill their cancerous cells.

The research study procedures include screening for eligibility, study treatment, including evaluations and follow up visits, blood collections, echocardiograms, and radiologic imaging of tumors.

It is expected participants will receive treatment over a period of short-term (approx. 2 years) and then long-term follow-up of up to 15 years.

It is expected that about 21 people will take part in this research study.

This research study has received funding through an internal grant program.

ELIGIBILITY:
Inclusion Criteria:

* Safety Run In Arm and ARM 1: Recurrent GBM, EGFRvIII mutant

  * Participants must have histologically confirmed recurrent GBM or molecular features of GBM with presence of EGFRvIII mutation detected at initial diagnosis. MGMT methylated, unmethylated, or unknown is allowed.
  * Participants must be at first progression or recurrence and plan is for biopsy or surgical debulking. Participants must have at least received prior radiation. Prior temozolomide is not required if the participant is MGMT unmethylated.

Participants must be 2 weeks from prior alkylating therapy or immunotherapy and ≥ 5 half-lives from another investigational agent before proceeding with collection or treatment. No washout is required from radiation since participants will need histological confirmation of recurrence to participate.

* ARM 2: Newly Diagnosed GBM, EGFRvIII mutant (will only open once safety is confirmed in Arms 1 and 3)

  * Participants must have histologically confirmed newly diagnosed GBM with presence of EGFRvIII mutation and their tumors must be MGMT unmethylated.
  * Treatment planned with involved field radiation alone without concomitant or sequential temozolomide.
* ARM 3: Recurrent GBM, EGFRvIII negative

  * Participants must have histologically confirmed recurrent GBM with EGFR amplification but no EGFRvIII mutation based on initial diagnostic tissue.
  * Participants must be at first recurrence and plan is for biopsy or surgical debulking. Participants must have at least received prior radiation. Prior temozolomide is not required if the participant is MGMT unmethylated.

Participants must be 2 weeks from prior alkylating therapy or immunotherapy and ≥ 5 half-lives from another investigational agent. No washout is required from radiation since participants will need histological confirmation of recurrence to participate.

* ARM 1: Recurrent GBM, EGFRvIII mutant and ARM 3: Recurrent GBM, EGFRvIII negative:

  * Must be at least 3 months from completion of radiation or evidence of progression is outside the high dose radiation field.
* Safety Run-In Arm and ARM 1: Recurrent GBM, EGFRvIII mutant and ARM 3: Recurrent GBM, EGFRvIII negative:

  * Participants must have measurable disease, defined as at least one lesion ≥10 mm (≥1 cm) with MRI. See Section 11 (Measurement of Effect) for the evaluation of measurable disease.
* ALL ARMS:

  * Patients cannot have posterior fossa or intramedullary spine-only disease. Leptomeningeal disease is allowed anywhere in the neuroaxis. See Section 11 (Measurement of Effect) for the evaluation of measurable disease.
  * Resolution of AEs from any prior systemic anticancer therapy or radiotherapy to Grade 1 or baseline (except Grade 2 alopecia and Grade 2 sensory neuropathy)
  * Medically able and willing to undergo placement of an Ommaya reservoir.
  * Steroid dose anticipated to be ≤ 4 mg of dexamethasone a day or equivalent at time of first CAR-v3-TEAM-E infusion.
  * Age ≥18 years
  * Karnofsky ≥60%
  * Must be able to undergo an MRI with contrast.
  * Life expectancy of greater than 3 months.
  * Participants must have adequate organ and marrow function as defined below:

    * Absolute neutrophil count ≥1,000/mcL
    * Platelets ≥80,000/mcL
    * Total bilirubin ≤ institutional upper limit of normal (ULN); For patients with Gilbert's syndrome, total bilirubin can be ≤ 3xULN.
    * AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN
    * CrCl ≥ 60 mL/min
  * Participant has no prior history of malignancy, unless the subject has been free of the disease for ≥5 years with the exception of the following noninvasive malignancies:

    * Basal cell carcinoma of the skin
    * Squamous cell carcinoma of the skin
    * Carcinoma in situ of the cervix
    * Carcinoma in situ of the breast
    * Incidental histologic finding of prostate cancer (T1a or T1b) or prostate cancer that is curative
  * Left ventricular ejection fraction >50% as determined by TTE.
  * The effects of CARv3-TEAM-E on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of CARv3-TEAM-E administration.
  * Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Intraparenchymal posterior fossa disease
* Intramedullary spinal disease as the only site of disease.
* Prior EGFRvIII targeted therapies.
* Prior bevacizumab treatment.
* Treatment with an any prior gene-therapy or gene-modified cellular therapy.
* Patients with a VP shunt or patients needing a shunt in the immediate future are excluded from participating
* Ongoing treatment with chronic immunosuppressants (e.g., cyclosporine or systemic steroids above physiologic dosing). Intermittent topical, inhaled, or intranasal corticosteroids are allowed
* Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia.
* Participants who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CARv3-TEAM-E (ex. cetuximab).
* Participants with uncontrolled intercurrent illness.
* Human immunodeficiency virus (HIV)-infected participants are not eligible.
* Participants with evidence of chronic hepatitis B virus (HBV) infection or active hepatitis C virus (HCV) infection are not eligible.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with CARv3-TEAM-E , breastfeeding should be discontinued if the mother is treated with CARv3-TEAM-E.
* For Arm 2, prior to CARv3-TEAM-E Infusion, the following criteria should be confirmed in addition to the relevant criteria above:

  * Participants must have completed 75% of the planned 6 weeks of involved field radiation without temozolomide
  * Tumor location and size criteria as in 3.1.7 above.
  * Prior cancer directed therapy other than radiation is not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | From Day 0 to 2 years post-treatment
  Defined as the incidence of ≥ Grade 3-4 adverse events related to CARv3-TEAM-E.
Number of Dose-Limiting Toxicities (DLTs) | up to 6 months
  Defined as any related toxicity experienced by run-in cohort of CTCAE v5 grade ≥ 4 Adverse Event

SECONDARY OUTCOMES:
Proportion of Participants with One Infusion | up to 6 months
  The study will be deemed feasible if the proportion of participants enrolled that go on to receive at least one infusion of CARv3-TEAM-E cells is 60% or greater. Applies to participants in run-in cohort and Arms 1 and 3.
Overall Response Rate | Day 0 to 2 years post-treatment
  Defined as the best response recorded from the start of treatment until disease progression/recurrence and evaluated using the Response Assessment in Neuro-Oncology Criteria (RANO).
Overall Survival Rate | From Day 0 to 2 years post-treatment
  Defined as the time from registration to death due to any cause.
Progression Free Survival (PFS) | Registration to 2 years post-treatment
  Defined as the time from registration to the earlier of progression or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: William Curry, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Choi BD, Gerstner ER, Frigault MJ, Leick MB, Mount CW, Balaj L, Nikiforow S, Carter BS, Curry WT, Gallagher K, Maus MV. Intraventricular CARv3-TEAM-E T Cells in Recurrent Glioblastoma. N Engl J Med. 2024 Apr 11;390(14):1290-1298. doi: 10.1056/NEJMoa2314390. Epub 2024 Mar 13. PMID 38477966